CLINICAL TRIAL: NCT07047482
Title: Clinicopathological Value of p16 Expression in Colorectal Carcinoma: An Immunohistochemical Study.
Brief Title: Clinicopathological Value of p16 Expression in Colorectal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherry Raouf Azmy, Demonstrator of pathology, Sohag University
Other Study IDs: Soh-Med--25-6-2MS
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Carcinoma
Keywords: p16 Expression; Colorectal Carcinoma; Immunohistochemical study
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fifty (50) cases of colorectal cancer will be performed from archieved formalin-fixed, paraffin-embedded tissue blocks referred to Pathology Department, Sohag University Hospitals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Fifty (50) cases of colorectal cancer will be performed from archieved formalin-fixed, paraffin-embedded tissue blocks referred to Pathology Department, Sohag University Hospitals.
  Interventions: Biological: Immunohistochemical staining

INTERVENTIONS:
Biological: Immunohistochemical staining — Immunohistochemical staining of paraffin embedded blocks of colorectal carcinoma tissues by p16 monoclonal antibodies to be evaluated with the positivity, intensity and distribution of the detected stain.

SUMMARY:
Evaluation of the immunohistochemical expression of p16 in colorectal carcinoma and correlate its expression to different clinical and pathological parameters as patients' ages, sexes, tumor location, histopathological phenotype, status of nodal involvement, perineural and lymphovascular invasion.

DETAILED DESCRIPTION:
Colorectal Carcinoma is very common nowadays, with increasing need for further research.

p16 is tumor suppressor gene with a vital rule ; inactivation of p16 leads to tumor formation and progression.

50 Specimens will be collected from Pathology Department of Sohag University Hospital. Sufficient clinical and histopathological data will be attached for each case.

The previously processed formalin-fixed, paraffin-embedded tissue blocks will be used to get Hematoxylin & Eosin stained sections to confirm the diagnosis and to detect the histopathological type, grade and stage of each tumor.

Another sliced tissue sections will be immunohistochemically stained with p16 monoclonal antibodies to be evaluated with the positivity, intensity and distribution of the detected stain.

ELIGIBILITY:
Inclusion Criteria:

1. Specimens from patients with colorectal cancer.
2. Tissue blocks with sufficient material.
3. Specimens with sufficient clinical data.

Exclusion Criteria:

1. Tissue blocks with insufficient, destroyed or necrotic material.
2. Specimens with insufficient clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifty (50) cases of colorectal cancer will be performed from archieved formalin-fixed, paraffin-embedded tissue blocks referred to Pathology Department, Sohag University Hospitals.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of p16 Expression in Colorectal Carcinoma. | 6 months
  Immunohistochemical staining of Colorectal tissues by p16 monoclonal antibody

SECONDARY OUTCOMES:
Correlation of p16 expression to different clinical and pathological parameters | 6 months
  Correlation of p16 expression to different clinical and pathological parameters as patients' ages, sexes, tumor location, histopathological phenotype, status of nodal involvement, perineural and lymphovascular invasion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag, Recruiting, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet